CLINICAL TRIAL: NCT00084318
Title: A Phase II Randomized Trial Of Surgery Followed By Chemoradiotherapy Plus Cetuximab For Advanced Squamous Cell Carcinoma Of The Head and Neck
Brief Title: Adjuvant Cetuximab and Chemoradiotherapy Using Either Cisplatin or Docetaxel in Treating Patients With Resected Stage III or Stage IV Squamous Cell Carcinoma or Lymphoepithelioma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0234; CDR0000360850; NCT00414674 (obsolete NCT alias)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2016-12

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III lymphoepithelioma of the oropharynx; stage IV lymphoepithelioma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT + cisplatin + cetuximab (Experimental): Loading dose of cetuximab followed by radiation therapy with weekly cisplatin and cetuximab.
  Interventions: Biological: cetuximab; Drug: cisplatin; Radiation: radiation therapy
- RT + docetaxel + cetuximab (Experimental): Loading dose of cetuximab followed by radiation therapy (RT) with weekly docetaxel and cetuximab.
  Interventions: Biological: cetuximab; Drug: docetaxel; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab — 400 mg/m^2 intravenously over 120 minutes on day 1 (week 1) followed by 250 mg/m^2 intravenously over 60 minutes in weeks 2 through 7.
Drug: cisplatin — 30 mg/m^2 intravenously infused over over 60 minutes in weeks 2 through 7.
  Arms: RT + cisplatin + cetuximab
Drug: docetaxel — 15 mg/m^2 intravenously infused over 30 minutes in weeks 2 through 7.
  Arms: RT + docetaxel + cetuximab
Radiation: radiation therapy — 60 Gy (2 Gy once a day, 5 times a week)

SUMMARY:
RATIONALE: Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as cisplatin and docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Cisplatin and docetaxel may make the tumor cells more sensitive to radiation therapy. Combining a monoclonal antibody with chemoradiotherapy and giving them after surgery may kill any remaining tumor cells.

PURPOSE: This randomized phase II trial is studying adjuvant cetuximab given together with chemoradiotherapy using cisplatin to see how well it works compared to adjuvant cetuximab given together with chemoradiotherapy using docetaxel in treating patients with resected stage III or stage IV squamous cell carcinoma (cancer) or lymphoepithelioma of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare disease-free survival of patients with resected stage III or IV squamous cell carcinoma or lymphoepithelioma of the head and neck treated with adjuvant cetuximab in combination with chemoradiotherapy comprising docetaxel vs cisplatin.

Secondary

* Compare the safety and efficacy of these regimens in these patients.
* Compare locoregional control and overall survival rates in patients treated with these regimens.
* Correlate epidermal growth factor receptor (total and phosphorylated), pMAPK, pAKT, Stat-3, Ki-67, cyclo-oxygenase-2, and cyclin B1 expression with outcome in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to Zubrod performance status (0 vs 1), risk category (positive margins vs high risk [i.e., ≥ 2 positive nodes or extracapsular nodal extension]) and use of intensity-modulated radiotherapy (no vs yes). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cetuximab IV over 2 hours on day 1 (week 1). Patients then receive cetuximab IV over 1 hour and cisplatin IV over 1 hour before radiotherapy on days 8, 15, 22, 29, 36, and 43 (weeks 2-7). Patients undergo radiotherapy once daily, 5 days a week, beginning on day 8 for a total of 6 weeks (weeks 2-7).
* Arm II: Patients receive cetuximab and undergo radiotherapy as in arm I. Patients also receive docetaxel IV over 30 minutes before radiotherapy on days 8, 15, 22, 29, 36, and 43 (weeks 2-7).

Treatment in both arms continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 230 patients (115 per treatment arm) will be accrued for this study within approximately 29 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck meeting the following criteria:

  * Site of tumor origin in the oral cavity, oropharynx, larynx, or hypopharynx (excluding lip, nasopharynx, or sinuses)
  * Gross total resection must be completed within 7 weeks of randomization, with pathology demonstrating one or more of the following risk factors:

    * Histologic extracapsular nodal extension
    * Histologic involvement of ≥ 2 regional lymph nodes
    * Invasive cancer seen on microscopic evaluation of the resection margin, with no evidence of gross tumor residual.
    * Tonsillar cancer patients who undergo transoral excision of all gross tumor are eligible provided extracapsular nodal extension or involvement of ≥ 2 regional lymph nodes is histologically confirmed
  * American Joint Committee on Cancer (AJCC) pathological stage III or IV
* No evidence of distant metastases
* No synchronous or concurrent head and neck primary tumors

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 8.0 g/dL

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT), and alkaline phosphatase meeting 1 of the following parameters:

  * Alkaline phosphatase ≤ ULN AND AST or ALT ≤ 5 times ULN
  * Alkaline phosphatase ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * Alkaline phosphatase ≤ 5 times ULN AND AST or ALT ≤ ULN

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No unstable angina
* No uncontrolled hypertension
* No myocardial infarction within the past 6 months (unless successfully treated with coronary artery bypass surgery or percutaneous transluminal coronary angioplasty)
* No uncontrolled arrhythmia
* No congestive heart failure
* No more than 2 heart-related hospitalizations within the past year
* No other active cardiac disease

Pulmonary

* No more than 2 hospitalizations for chronic obstructive pulmonary disease within the past year

Neurologic

* No pre-existing peripheral neuropathy ≥ grade 2
* No uncontrolled seizure disorder
* No active neurological disease

Other

* No prior severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No other invasive malignancy within the past 3 years except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior anti-epidermal growth factor receptor antibody therapy

Chemotherapy

* More than 3 years since prior cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior head and neck radiotherapy

Surgery

* See Disease Characteristics

Other

* No prior tyrosine kinase inhibitor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2004-04; Primary Completion 2009-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Harari, MD, Principal Investigator — University of Wisconsin, Madison; Merrill S. Kies, MD, Study Chair — M.D. Anderson Cancer Center; Jeffrey N. Myers, MD, PhD, FACS, Study Chair — M.D. Anderson Cancer Center
Locations (160):
- United States (160):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Osborn, Scottsdale, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Torrance Memorial Medical Center, Torrance, California
  - Solano Radiation Oncology Center, Vacaville, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Hospital of Saint Raphael, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lynn Regional Cancer Center at Boca Raton Community Hospital - Main Center, Boca Raton, Florida
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - John D. Cronin Cancer Center, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Tulane Cancer Center, Alexandria, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Long Island College Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Mercy Cancer Institute at Mercy Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin

REFERENCES:
- [Result] Harari PM, Harris J, Kies MS, et al.: Phase II randomized trial of surgery followed by chemoradiation plus cetuximab for high-risk squamous cell carcinoma of the head and neck (RTOG 0234). [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-22, S13, 2007.
- [Result] Harari PM, Harris J, Kies MS, Myers JN, Jordan RC, Gillison ML, Foote RL, Machtay M, Rotman M, Khuntia D, Straube W, Zhang Q, Ang K. Postoperative chemoradiotherapy and cetuximab for high-risk squamous cell carcinoma of the head and neck: Radiation Therapy Oncology Group RTOG-0234. J Clin Oncol. 2014 Aug 10;32(23):2486-95. doi: 10.1200/JCO.2013.53.9163. Epub 2014 Jul 7. PMID 25002723

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RT + Cisplatin + Cetuximab | RT + Docetaxel + Cetuximab
Started | 119 | 119
Completed | 97 (Subjects with data available for the primary analysis are considered to have completed the study.) | 106 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 22 | 13
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Protocol Violation | 15 | 11
Not completed — No protocol treatment | 2 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients who started protocol treatment and did not withdraw consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | RT + Cisplatin + Cetuximab | RT + Docetaxel + Cetuximab | Total
Number analyzed (Participants) | 97 | 106 | 203
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 80] | 55 [21 to 79] | 56 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 32 | 52
  Male | 77 | 74 | 151

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Two-year rates are shown (Kaplan-Meier estimates). Disease-free survival is defined as the time from randomization to local, regional, or distant progression, second primary, or death (event) or last follow-up (censored). Response criteria as follows: No evidence of disease (NED): All patients must have no measurable tumor following surgery; Local-Regional Relapse: Recurrent cancer in the tumor bed and/or neck not clearly attributable to a second primary neoplasm; biopsy confirmation is necessary; Distant Relapse: Clear evidence of distant metastases (lung, bone, brain, etc.); Biopsy is recommended where possible. A solitary lung mass/nodule is considered a second primary neoplasm unless proven otherwise.
Time Frame: From randomization to 2 years
Population: Eligible patients who started protocol treatment and did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin + Cetuximab | RT + Docetaxel + Cetuximab
Number analyzed (Participants) | 97 | 106
percentage of participants | 57.3 [47.4 to 67.2] | 65.9 [56.9 to 75]
Statistical Analysis 1: Comparison: RT + Cisplatin + Cetuximab; Using the method of Dixon and Simon, 104 analyzable patients per arm were needed to detect a ≥ 33 reduction in the hazard rate for disease-free survival compared to historical control data (the chemoradiation arm of study RTOG-9501/NCT00002670) with 80% power and one-sided log-rank test at the 0.05 level. Two-year rates were estimated by the Kaplan-Meier method. [RTOG = Radiation Therapy Oncology Group]; Test type: Superiority or Other; p = 0.05, Log Rank; Historical control data (RTOG-9501/NCT00002670): n=202, two-year disease-free survival rate of 54.8% (47.9% to 61.7%); Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.54 to 1.06]
Statistical Analysis 2: Comparison: RT + Docetaxel + Cetuximab; Using the method of Dixon and Simon, 104 analyzable patients per arm were needed to detect a ≥ 33 reduction in the hazard rate for disease-free survival compared to historical control data (the chemoradiation arm of study RTOG-9501/NCT00002670) with 80% power and one-sided log-rank test at the 0.05 level. Two-year rates were estimated by the Kaplan-Meier method; Test type: Superiority or Other; p = 0.01, Log Rank; Historical control data (RTOG-9501/NCT00002670): n=202, two-year disease-free survival rate of 54.8% (47.9% to 61.7%); Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.50 to 0.96]

2. Secondary Outcome: Overall Survival
Description: Two-year rates are shown (Kaplan-Meier estimates). Overall survival is defined as the time from randomization to death (event) or last follow-up (censored).
Time Frame: From randomization to 2 years
Population: Eligible patients who started protocol treatment and did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin + Cetuximab | RT + Docetaxel + Cetuximab
Number analyzed (Participants) | 97 | 106
percentage of participants | 68.8 [59.5 to 78] | 79.2 [71.4 to 86.9]
Statistical Analysis 1: Comparison: RT + Cisplatin + Cetuximab; Two-year rates were estimated by the Kaplan-Meier method. RTOG 0234 results were compared to historical control data (the chemoradiation arm of study RTOG-9501/NCT00002670) by 1-sided log-rank test. Hazard ratios were estimated by Cox model. [RTOG = Radiation Therapy Oncology Group]; Test type: Superiority or Other; p = 0.04, Log Rank; Historical control data (RTOG-9501/NCT00002670): n=202, two-year survival rate of 64.7% (58.1% to 71.3%); Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.5 to 1.03] — Reference arm = historical control
Statistical Analysis 2: Comparison: RT + Docetaxel + Cetuximab; Two-year rates were estimated by the Kaplan-Meier method. RTOG 0234 results were compared to historical control data (the chemoradiation arm of study RTOG-9501/NCT00002670) by 1-sided log-rank test. Hazard ratios were estimated by Cox model; Test type: Superiority or Other; p = 0.001, Log Rank; Historical control data (RTOG-9501/NCT00002670): n=202, two-year survival rate of 64.7% (58.1% to 71.3%); Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.39 to 0.82] — Reference arm = historical control

3. Secondary Outcome: Treatment Tolerance
Description: Tolerability was defined as having received 90% of the radiation dose, 95% of the cetuximab loading dose, and at least 4 weeks of cetuximab and cisplatin or docetaxel at doses 95% of the protocol prescription. The percentage of patients determined to be tolerant of treatment are shown.
Time Frame: From start of treatment to end of treatment (protocol treatment lasts seven weeks).
Population: Eligible patients who started protocol treatment and did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RT+Cisplatin+Cetuximab: Loading dose of cetuximab followed by radiation therapy with weekly cisplatin and cetuximab.
- RT+Docetaxel+Cetuximab: Loading dose of cetuximab followed by radiation therapy (RT) with weekly docetaxel and cetuximab.
Arm/Group | RT+Cisplatin+Cetuximab | RT+Docetaxel+Cetuximab
Number analyzed (Participants) | 97 | 106
percentage of participants | 80.4 [72.5 to 88.3] | 84.9 [78.1 to 91.7]

4. Secondary Outcome: Frequency of Toxicity (Grade 5 and Acute Non-hematologic Grade 4)
Description: Each regimen was monitored for excessive acute toxicity (defined as nonhematologic grade 4 toxicity within 90 days of the start of radiation or any grade 5 toxicity). The target rate was based on the observed rate from RTOG-9501/NCT00002670 of 15%. The unacceptable rate was >30%. [RTOG = Radiation Therapy Oncology Group]
Time Frame: From start of treatment to last follow-up. Analysis occurs at the time of the primary analysis.
Population: Eligible patients who started protocol treatment and did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT+Cisplatin+Cetuximab | RT+Docetaxel+Cetuximab
Number analyzed (Participants) | 97 | 106
percentage of participants | 9.3 [3.5 to 15.1] | 12.3 [6.0 to 18.5]

5. Secondary Outcome: Frequency of Other Acute and Late Toxicity
Description: Maximum grade toxicity that is definitely, probably, or possibly related to protocol treatment.
Time Frame: From start of treatment to last follow-up. Analysis occurs at the time of the primary endpoint analysis.
Population: Eligible patients who started protocol treatment and did not withdraw consent
Measure: Number; unit: percentage of participants
Arm/Group | RT+Cisplatin+Cetuximab | RT+Docetaxel+Cetuximab
Number analyzed (Participants) | 97 | 106
percentage of participants
  Grade 1 | 1.0 | 0.0
  Grade 2 | 10.3 | 9.4
  Grade 3 | 74.2 | 73.6
  Grade 4 | 14.4 | 16.0
  Grade 5 | 0.0 | 0.9

6. Secondary Outcome: Local-regional Control
Description: Two-year rate is shown (cumulative incidence estimate). Local-regional failure is defined as the time from randomization to local-regional recurrence (event), death (competing risk), or last follow-up (censored).
Time Frame: From randomization to 2 years
Population: Eligible patients who started protocol treatment and did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cisplatin + Cetuximab | RT + Docetaxel + Cetuximab
Number analyzed (Participants) | 97 | 106
percentage of participants | 19.8 [11.8 to 27.8] | 18.9 [13.4 to 24.3]
Statistical Analysis 1: Comparison: RT + Cisplatin + Cetuximab; Two-year failure rates were estimated by the cumulative incidence method. RTOG 0234 results were compared to historical control data (the chemoradiation arm of study RTOG-9501/NCT00002670) by 1-sided Gray's test. Hazard ratios were estimated by Cox model. [RTOG = Radiation Therapy Oncology Group]; Test type: Superiority or Other; p = 0.66, Gray's test; Historical control data (RTOG-9501/NCT00002670): n=202, two-year failure rate of 19.9% (12.2% to 27.5%); Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.63 to 1.76] — Reference arm = historical control
Statistical Analysis 2: Comparison: RT + Docetaxel + Cetuximab; Two-year failure rates were estimated by the cumulative incidence method. RTOG 0234 results were compared to historical control data (the chemoradiation arm of study RTOG-9501/NCT00002670) by 1-sided Gray's test. Hazard ratios were estimated by Cox model; Test type: Superiority or Other; p = 0.86, Gray's test; Historical control data (RTOG-9501/NCT00002670): n=202, two-year failure rate of 19.9% (12.2% to 27.5%); Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.72 to 1.87] — Reference arm = historical control

7. Secondary Outcome: Correlation of EGFR (Total and Phosphorylated) pMAPK, pAKT, Stat-3, KI-67, COX-2, and Cyclin B1 Expression With Local-regional Control, and Overall and Disease-free Survival
Time Frame: From randomization to two years
Population: Effective and reliable assessment of nuclear expression of these receptors was not achieved and therefore no data was available for analysis.
Arm/Group | RT + Cisplatin + Cetuximab | RT + Docetaxel + Cetuximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events.
Arm/Group | RT+Cisplatin+Cetuximab | RT+Docetaxel+Cetuximab
Serious Adverse Events (participants affected / at risk) | 42/97 | 56/106
Other Adverse Events (participants affected / at risk) | 97/97 | 105/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RT+Cisplatin+Cetuximab (N=97) | RT+Docetaxel+Cetuximab (N=106)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0
Hemoglobin (Blood and lymphatic system disorders) | 6 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac general - Other (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 2
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 1
Acquired tracheo-esophageal fistula (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhea NOS (Gastrointestinal disorders) | 3 | 4
Dry mouth (Gastrointestinal disorders) | 9 | 13
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 10 | 11
Esophageal stenosis acquired (Gastrointestinal disorders) | 0 | 1
Esophagitis NOS (Gastrointestinal disorders) | 1 | 2
Fistula, GI: Oral cavity (Gastrointestinal disorders) | 0 | 2
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 2
Mucositis/stomatitis (clinical exam): Large bowel (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 7
Oral pain (Gastrointestinal disorders) | 2 | 5
Radiation mucositis (Gastrointestinal disorders) | 10 | 12
Salivary gland disorder NOS (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 8
Vomiting NOS (Gastrointestinal disorders) | 5 | 8
Constitutional Symptoms - Other (General disorders) | 0 | 1
Edema: head and neck (General disorders) | 1 | 4
Fatigue (General disorders) | 5 | 4
Pain - Other (General disorders) | 1 | 4
Pyrexia (General disorders) | 2 | 10
Rigors (General disorders) | 0 | 4
Hypersensitivity NOS (Immune system disorders) | 2 | 4
Bladder infection NOS (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 1 | 3
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Bladder (urinary) (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Middle ear (otitis media) (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Sinus (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Skin (cellulitis) (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Blood (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Catheter-related (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Neck NOS (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Salivary gland (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1 | 0
Infection with unknown ANC: Neck NOS (Infections and infestations) | 0 | 1
Infection with unknown ANC: Pharynx (Infections and infestations) | 1 | 0
Infection with unknown ANC: Trachea (Infections and infestations) | 1 | 0
Infectous meningitis (Infections and infestations) | 0 | 1
Opportunisitic infection (Infections and infestations) | 0 | 1
Pneumonia NOS (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 1 | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 2 | 6
Radiation recall syndrome (Injury, poisoning and procedural complications) | 3 | 4
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 2
Leukopenia NOS (Investigations) | 5 | 0
Lymphopenia (Investigations) | 5 | 2
Neutrophil count (Investigations) | 5 | 0
Platelet count decreased (Investigations) | 3 | 0
Weight decreased (Investigations) | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 8 | 6
Hyperglycemia NOS (Metabolism and nutrition disorders) | 2 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycemia NOS (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal/soft tissue - Other (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 3
Ataxia (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 3 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Mental status changes (Nervous system disorders) | 0 | 1
Neurology - Other (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Renal failure NOS (Renal and urinary disorders) | 1 | 2
Renal/genitourinary - Other (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Mucositis/stomatitis (clinical exam): Pharynx (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Mucositis/stomatitis (functional/symptomatic): Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne NOS (Skin and subcutaneous tissue disorders) | 2 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 4 | 2
Dermatology/skin - Other (Skin and subcutaneous tissue disorders) | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Fat atrophy NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pain: Scalp (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction NOS (Skin and subcutaneous tissue disorders) | 1 | 1
Skin fibrosis (Skin and subcutaneous tissue disorders) | 3 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RT+Cisplatin+Cetuximab (N=97) | RT+Docetaxel+Cetuximab (N=106)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 6 | 5
Hemoglobin (Blood and lymphatic system disorders) | 57 | 55
Auditory/ear - Other (Ear and labyrinth disorders) | 6 | 5
Hearing impaired (Ear and labyrinth disorders) | 3 | 10
Tinnitus (Ear and labyrinth disorders) | 5 | 6
Hypothyroidism (Endocrine disorders) | 10 | 15
Abdominal pain NOS (Gastrointestinal disorders) | 6 | 7
Constipation (Gastrointestinal disorders) | 26 | 35
Diarrhea NOS (Gastrointestinal disorders) | 23 | 23
Dry mouth (Gastrointestinal disorders) | 79 | 85
Dyspepsia (Gastrointestinal disorders) | 7 | 13
Dysphagia (Gastrointestinal disorders) | 74 | 86
Esophageal stenosis acquired (Gastrointestinal disorders) | 7 | 8
Esophagitis NOS (Gastrointestinal disorders) | 9 | 17
Gastrointestinal - Other (Gastrointestinal disorders) | 10 | 12
Nausea (Gastrointestinal disorders) | 53 | 49
Oral pain (Gastrointestinal disorders) | 29 | 42
Radiation mucositis (Gastrointestinal disorders) | 55 | 65
Salivary gland disorder NOS (Gastrointestinal disorders) | 29 | 36
Stomatitis (Gastrointestinal disorders) | 21 | 34
Tooth disorder NOS (Gastrointestinal disorders) | 6 | 6
Vomiting NOS (Gastrointestinal disorders) | 33 | 27
Edema: head and neck (General disorders) | 24 | 27
Facial pain (General disorders) | 3 | 7
Fatigue (General disorders) | 76 | 83
Pain - Other (General disorders) | 12 | 9
Pyrexia (General disorders) | 16 | 16
Rigors (General disorders) | 7 | 11
Gingival infection (Infections and infestations) | 6 | 3
Infection - Other (Infections and infestations) | 10 | 8
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 39 | 47
Radiation recall syndrome (Injury, poisoning and procedural complications) | 29 | 19
Alanine aminotransferase increased (Investigations) | 8 | 16
Aspartate aminotransferase increased (Investigations) | 17 | 24
Blood alkaline phosphatase increased (Investigations) | 7 | 16
Blood bilirubin increased (Investigations) | 7 | 8
Blood creatinine increased (Investigations) | 5 | 5
Leukopenia NOS (Investigations) | 51 | 29
Lymphopenia (Investigations) | 20 | 24
Metabolic/laboratory - Other (Investigations) | 7 | 11
Neutrophil count (Investigations) | 20 | 6
Platelet count decreased (Investigations) | 17 | 10
Weight decreased (Investigations) | 51 | 43
Anorexia (Metabolism and nutrition disorders) | 51 | 41
Dehydration (Metabolism and nutrition disorders) | 28 | 12
Hypercalcemia (Metabolism and nutrition disorders) | 9 | 4
Hyperglycemia NOS (Metabolism and nutrition disorders) | 40 | 30
Hyperkalemia (Metabolism and nutrition disorders) | 13 | 9
Hypermagnesemia (Metabolism and nutrition disorders) | 4 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 22 | 29
Hypocalcemia (Metabolism and nutrition disorders) | 16 | 20
Hypokalemia (Metabolism and nutrition disorders) | 19 | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 24 | 10
Hyponatremia (Metabolism and nutrition disorders) | 38 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Fibrosis-cosmesis (Musculoskeletal and connective tissue disorders) | 7 | 11
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 11 | 20
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal/soft tissue - Other (Musculoskeletal and connective tissue disorders) | 5 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 20 | 16
Trismus (Musculoskeletal and connective tissue disorders) | 17 | 24
Dizziness (Nervous system disorders) | 16 | 5
Dysgeusia (Nervous system disorders) | 53 | 52
Headache (Nervous system disorders) | 31 | 28
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 12
Anxiety (Psychiatric disorders) | 9 | 8
Depression (Psychiatric disorders) | 14 | 13
Insomnia (Psychiatric disorders) | 12 | 19
Aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 25
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Laryngitis NOS (Respiratory, thoracic and mediastinal disorders) | 25 | 28
Mucositis/stomatitis (clinical exam): Pharynx (Respiratory, thoracic and mediastinal disorders) | 13 | 4
Mucositis/stomatitis (functional/symptomatic): Pharynx (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 18
Acne NOS (Skin and subcutaneous tissue disorders) | 60 | 57
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 22
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 23 | 33
Dermatology/skin - Other (Skin and subcutaneous tissue disorders) | 12 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 15
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 13
Skin fibrosis (Skin and subcutaneous tissue disorders) | 30 | 37
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 23 | 20
Sweating increased (Skin and subcutaneous tissue disorders) | 1 | 6
Telangiectasia (Skin and subcutaneous tissue disorders) | 6 | 15
Hypotension NOS (Vascular disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.